CLINICAL TRIAL: NCT04367792
Title: Pathology and Pathogenesis of Cardiac Injury in COVID-19 Infections in Humans
Brief Title: Cardiac Injury in COVID-19: a Pathology Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: CVPath Institute Inc. Renu Virmani, Aloke Finn (Unknown); A.O. Ospedale Papa Giovanni XXIII, Anatomia Patologica, Dr Andrea Gianatti, co-PI (Unknown)
Responsible Party: Principal Investigator, GGuagliumi, MD Cardiologist, A.O. Ospedale Papa Giovanni XXIII
Other Study IDs: 56/20
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: COVID-19
Keywords: Covid-19; Infectious disease; Health care; Heart disease; Viruses; Myocarditis; Pathology
MeSH Terms: conditions — COVID-19; Communicable Diseases; Heart Diseases; Virus Diseases; Myocarditis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients died with Covid-19 disease: Sample of patients died with Covid-19 disease and pulmonary disease
- Patients died with Covid-19 and cardiovascular disease: Sample of patients died with Covid-19 disease and pulmonary disease with clear cardiovascular involvement
- Patient died with myocarditis: Sample of patient died with different types of myocarditis without Covid-19 disease. These samples are used as control and are part of database of previously collected samples of CVPath Institute Inc.

SUMMARY:
The primary goal of the study is to conduct the first systematic cardiac autopsy study in 60 patients dying from COVID-19 to understand the pathology and pathogenesis of cardiac injury in patients with COVID-19, with/without cardiovascular comorbidities. Such data is essential for understanding rate of involvement, type of involvement and degree of injury in patients contracting the disease.

DETAILED DESCRIPTION:
Since Dec 2019, coronavirus disease 2019 (COVID-19) caused by the severe acute respiratory syndrome coronavirus 2(SARS-CoV-2) has resulted in considerable morbidity and mortality throughout the world. On April 21 2020, Italy and US have registered over 187,000 and 855,000 cases of confirmed COVID-19 disease respectively, with one of the highest death rates in the world, which stands at more than 25,000 individuals in Italy and 47,000 in US. Epidemiologic modeling from multiple groups indicate the scope of the problem, with a potential for over 200,000 deaths in the U.S. alone, with large percentage of the population infected. Mortality from COVID-19 is associated with the presence of severe respiratory illness, although recent studies indicate 20%-30% of patients have evidence of COVID-19 associated cardiac injury defined as decline in ejection fraction or troponin I elevation (1,2). Anecdotal evidence suggests the presence of abnormal EKG findings compatible with myocardial ischemia but whether this is from epicardial coronary thrombosis, myocarditis, or microvascular thrombosis remains uncertain although all have been postulated (3). Regardless, patients with cardiac injury have higher mortality than those without, and sudden cardiac death has been described in some of these patients (1). Two thirds of patients with cardiovascular history were more likely to develop cardiac complications (4). Isolated reports have described fulminant myocarditis in the setting of high viral load with autopsy findings consistent with inflammatory mononuclear infiltrates (5). However, no systematic autopsy studies of patients dying from COVID-19 have ever been conducted. The Papa Giovanni XXIII Hospital, Bergamo had treated about 2000 patients with COVID-19 and performed systematic cardiac autopsies from a series of 60 patients who died or presented with/without a picture of cardiac injury and were COVID-19 positive. Detailed clinical data on all these patients are available.

Background Much about the pathogenesis of SARS-CoV-2 and the heart remains unknown. Angiotensin (AT) converting enzyme 2 (ACE2) is known as the cellular receptor for both SARS-CoV and SARS-CoV-2 but also as an endogenous counter- regulator of the renin-angiotensin system (RAS). ACE2 is ubiquitously expressed with the highest levels detected in the cardiovascular system (cardiomyocytes, cardiac fibroblasts, vascular smooth muscle cells and endothelial cells) as well as gut, kidneys and lungs. In general, loss of ACE2 increases susceptibility to cardiovascular disease such as myocardial infarction and hypertension while gain of function ACE2 has shown protective roles in various models of cardiovascular disease (6). The bifunctional role of ACE2 as a receptor for SARS-COV-2 but also as a protective factor against cardiovascular disease means careful understanding of the role of ACE2 during SARS-CoV-2 is needed. In this proposal investigators will examine cardiac tissues from patients dying of COVID-19 and examine the effect of infection on the expression of ACE2 on various cardiac cells. Investigators will also evaluate and validate this hypothesized mechanism of viral entry by ACE2 and trans-membrane serine protease which promotes entry of SARS-COV-2 into cells through a separate mechanisms.

Study Aims:

1. Describe the cardiac pathological findings from series of 60 patients dying from COVID-19 using cardiac samples sent to CVPath Institution from Papa Giovanni XXIII Hospital, Bergamo, Italy to study the correlations between clinical risk factors and myocardial findings and difference from other viral myocarditis;
2. Understand the relationship between viral load in cardiac tissues and the extent of damage seen on myocardial histological sections; and
3. Co-localize the SARS-CoV-2 using RNAscope in situ hybridization, with its entry receptor ACE2 and serine protease TMPRSS2 (type II transmembrane serine protease) in different cell types found in the heart, such as endothelial, smooth muscle, myocardial, fibroblastic and inflammatory cells, to better understand the pathogenesis of the disease.

Methods:

The study was approved by ethical committee at Papa Giovanni XXIII Hospital and the CVPath Institute IRB (Institutional Review Board).

All specimens are fixed in 10% buffered formalin. Hearts will be shipped to CVPath in accordance with all international shipping regulations and U.S. CDC (Centers for Disease Control and Prevention) guidelines (www.cdc.gov/coronavirus/2019-ncov/hcp/guidance-postmortem specimens.html). The sample is given a unique identifier and the hearts are weighed after blood clots have been removed from the cavities, and the heart ventricles are sliced parallel to the posterior atrioventricular junction to determine absence of any necrosis or fibrosis. Pulmonary emboli and any right ventricular abnormalities are assessed to rule out any attributable cause of death. The heart is weighed and radiographed and if any calcification is observed the epicardial coronary arteries are removed intact away from the heart and segments decalcified according to the extent of calcification. The rest of the arteries are submitted for paraffin embedding at 3-4 mm intervals to rule out any significant atherosclerosis (75 % cross-sectional area stenosis) or any thrombosis.

In total six sections of myocardium (anterior, posterior, and lateral LV (left ventricle), ventricular septum, anterior and posterior wall of the right ventricle) are routinely taken transversely, embedded in paraffin, and stained with hematoxylin and eosin (H&E) for histologic evaluation. If specific pathology is observed, additional sections will be submitted to determine the etiology of the findings. Histologic examination is performed to rule out any infiltrative or inflammatory process or any myofiber disarray of the myocardium, intramyocardial small vessel disease of interstitial or focal fibrosis. Presence of any cardiomyopathic process will be ruled out by gross and histologic examination. If the post-mortem interval is short, transmission electron microscopic (TEM) examination will be performed to determine the presence of virus and the cell type harboring the virus.

Correlations with autopsy findings will be made with available anonymized clinical data including EKG, echocardiography and cardiac catheterization (where available). The cardiac pathological characteristics of COVID-19 will be compared to 60 viral myocarditis cases that have previously been collected in CVPath Registry. A RT-PCR (reverse transcription polymerase chain reaction) specifically designed for SARS-CoV-2 will be conducted on RNA extracted from myocardial samples to quantitate the amount of virus in myocardium for each sample. RNA samples will also be taken from coronary arteries as well. Calculated viral load will be correlated with the myocardial injury scores including myocardial necrosis, myocardial infarction, myocarditis, inflammatory cells numbers, type, etc.

RNAscope In-situ hybridization. In situ detection of SARS-CoV-2 with ACE2 and TMPRSS2 in endothelial (VE-cadherin), myocardial (Cx43 and Myh6), smooth muscle cell (SM22 alpha) and lymphocytes (CD3, CD4, CD8) will be performed using an RNAscope assay with RNAscope Probe-V-nCoV2019-S-sense and Probe-V-nCoV2019-S (Advanced Cell Diagnostics) following the manufacturer's protocols. Correlation will be made with specific cell types mentioned by dual immunofluorescence as previously described (7) .

This study will result in a greater understanding of the pathology of cardiac injury in patients with COVID-19. Doing so will open the door to develop new therapeutic options to treat these patients during an epidemic of unparalleled size and scope.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients at Papa Giovanni XXIII Hospital, Bergamo, forefront of the COVIT-19 pandemic in Italy
* COVID-19 positive patients who died with/without a picture of cardiac injury

Exclusion Criteria:

* COVID-19 negative patients who died

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Systematic cardiac autopsy study of at least 60 patients dying from COVID-19 in Italy to understand the pathology and pathogenesis of cardiac injury in patients with COVID-19. Correlations with autopsy findings will be made with available anonymized clinical data including EKG, echocardiography and cardiac catheterization (where available). The cardiac pathologlical characteristics of COVID-19 will be compared to 60 viral myocarditis cases that have previously been collected in CVPath Registry.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Cardiac pathological findings from series of 60 patients dying from COVID-19 disease | 1 year
  Describe the cardiac pathological findings from series of 60 patients dying from COVID-19 using cardiac samples sent to CVPath Institution from Papa Giovanni XXIII Hospital, Bergamo to study the correlations between clinical risk factors and myocardial findings and difference from other viral myocarditis
viral load in cardiac tissues and the extent of damage | 1 year
  Understand the relationship between viral load in cardiac tissues and the extent of damage seen on myocardial histological sections
Co-localize the SARS-CoV-2 using RNAscope in situ hybridization, with its entry receptor ACE2 and serine protease TMPRSS2 in different cell types found in the heart | 1 year
  Co-localize the SARS-CoV-2 using RNAscope in situ hybridization, with its entry receptor ACE2 and serine protease TMPRSS2 in different cell types found in the heart, such as endothelial, smooth muscle, myocardial, fibroblastic and inflammatory cells to better understand the pathogenesis of the disease.

SECONDARY OUTCOMES:
Multi-organ involvement obtained from hystological analyses of paraffine blocks from different organs (ie kidney, spleen, bowel,....) | 1 year
  Multi-organ involvement associated with cardiac injury (microvascular and cardiomyocyte). If specific pathology is observed, additional sections from different organs (ie kidney, spleen, bowel) will be requested and submitted in paraffin blocks to determine the etiology of the findings. Histologic examination is performed to rule out any infiltrative or inflammatory process or any myofiber disarray of the myocardium, intramyocardial small vessel disease, including microvascular thrombosis of interstitial or focal fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: CTC CLINICAL TRIAL CENTER, Study Chair — Clinical Trials Center - Ospedale Papa Giovanni XXIII Bergamo
Locations (1):
- ASST Ospedale Papa Giovanni XXIII, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shi S, Qin M, Shen B, Cai Y, Liu T, Yang F, Gong W, Liu X, Liang J, Zhao Q, Huang H, Yang B, Huang C. Association of Cardiac Injury With Mortality in Hospitalized Patients With COVID-19 in Wuhan, China. JAMA Cardiol. 2020 Jul 1;5(7):802-810. doi: 10.1001/jamacardio.2020.0950. PMID 32211816
- [Background] Guo T, Fan Y, Chen M, Wu X, Zhang L, He T, Wang H, Wan J, Wang X, Lu Z. Cardiovascular Implications of Fatal Outcomes of Patients With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):811-818. doi: 10.1001/jamacardio.2020.1017. PMID 32219356
- [Background] Madjid M, Safavi-Naeini P, Solomon SD, Vardeny O. Potential Effects of Coronaviruses on the Cardiovascular System: A Review. JAMA Cardiol. 2020 Jul 1;5(7):831-840. doi: 10.1001/jamacardio.2020.1286. PMID 32219363
- [Background] Chen T, Wu D, Chen H, Yan W, Yang D, Chen G, Ma K, Xu D, Yu H, Wang H, Wang T, Guo W, Chen J, Ding C, Zhang X, Huang J, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical characteristics of 113 deceased patients with coronavirus disease 2019: retrospective study. BMJ. 2020 Mar 26;368:m1091. doi: 10.1136/bmj.m1091. PMID 32217556
- [Background] Alhogbani T. Acute myocarditis associated with novel Middle east respiratory syndrome coronavirus. Ann Saudi Med. 2016 Jan-Feb;36(1):78-80. doi: 10.5144/0256-4947.2016.78. PMID 26922692
- [Background] Zhong J, Basu R, Guo D, Chow FL, Byrns S, Schuster M, Loibner H, Wang XH, Penninger JM, Kassiri Z, Oudit GY. Angiotensin-converting enzyme 2 suppresses pathological hypertrophy, myocardial fibrosis, and cardiac dysfunction. Circulation. 2010 Aug 17;122(7):717-28, 18 p following 728. doi: 10.1161/CIRCULATIONAHA.110.955369. Epub 2010 Aug 2. PMID 20679547
- [Background] Guo L, Akahori H, Harari E, Smith SL, Polavarapu R, Karmali V, Otsuka F, Gannon RL, Braumann RE, Dickinson MH, Gupta A, Jenkins AL, Lipinski MJ, Kim J, Chhour P, de Vries PS, Jinnouchi H, Kutys R, Mori H, Kutyna MD, Torii S, Sakamoto A, Choi CU, Cheng Q, Grove ML, Sawan MA, Zhang Y, Cao Y, Kolodgie FD, Cormode DP, Arking DE, Boerwinkle E, Morrison AC, Erdmann J, Sotoodehnia N, Virmani R, Finn AV. CD163+ macrophages promote angiogenesis and vascular permeability accompanied by inflammation in atherosclerosis. J Clin Invest. 2018 Mar 1;128(3):1106-1124. doi: 10.1172/JCI93025. Epub 2018 Feb 19. PMID 29457790